CLINICAL TRIAL: NCT01629342
Title: Standardized Physical Activities Measured by Accelerometers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hillerod Hospital, Denmark (Other)
Responsible Party: Principal Investigator, Anna Maria Strømmen, principal investigator, Hillerod Hospital, Denmark
Other Study IDs: H-1-2012-001
Record Dates: First submitted 2012-06-25; First posted 2012-06-27 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2012-06

CONDITIONS: Transient Ischemic Attack
MeSH Terms: conditions — Ischemic Attack, Transient

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Transient Ischemic Attack Patients: Patients discharged after a Transient Ischemic Attack
  Interventions: Behavioral: Standardized activities

INTERVENTIONS:
Behavioral: Standardized activities — All patients do each of the following standardized activities over a course of 2 days:
  * treadmill walking (5 minutes, 1 and 2km/h)
  * staircase walking (1 floor, normal pace)
  * cycling with fixed load (5 minutes)
  * standing up from sitting position and sitting down again (x5)
  * standing up from supine position
  * turning from left to right and back while lying in bed
  * raising outstretched arm 90° (x5, standing position)
  * eating (5 minutes, sitting position)
  * drinking a glass of water
  * sleeping (6 hours)

SUMMARY:
STANDARDIZED PHYSICAL ACTIVITIES MEASURED BY ACCELEROMETERS Background and aims: Physical activity may be assessed by several different methods. However, the use of accelerometers is the most direct method available for real-time measurements. The piezoelectric element of accelerometers records an electric voltage during movement which is then transcribed to Activity Counts (AC). Few studies have used Actical accelerometers to assess standardized physical activities and most of these were not applicable to patients in a hospital setting. No previous studies have applied Actical accelerometers to the wrists or ankles during standardized activities. The aim of this study is to record AC during different standardized activities frequently done by patients hospitalized for acute ischemic stroke.

Methods: Patients discharged since February 2012 after a transient ischemic attack have been invited to participate in the study scheduled for June-September 2012 (nexpected=25). All participants wear 5 accelerometers (Actical), one at each wrist and ankle and one over the hip. Standardized physical activities include:

* treadmill walking (5 minutes, 1 and 4km/h)
* staircase walking (1 floor, normal pace)
* cycling with fixed load (5 minutes)
* standing up from sitting position and sitting down again (x5)
* standing up from supine position
* turning from left to right and back while lying in bed
* raising outstretched arm 90° (x5, standing position)
* eating (5 minutes, sitting position)
* drinking a glass of water
* sleeping (6 hours)

ELIGIBILITY:
Inclusion Criteria:

* Previous Transient Ischemic Attack
* age > 18 years

Exclusion Criteria:

* pregnancy and lactation
* time limit of more than 2 days of standardized activities exceeded
* no informed consent
* disability when tested with Scandinavian Stroke Scale (score <58), National Institutes of Health Stroke Scale (score >0), modified Rankin Scale (score >0) and Barthels Index 100 (score <100)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients just prior discharge from Stoke Unit, Neurologic Department, Hillerød Hospital
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2012-06; Primary Completion 2012-09 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Activity | 2 days
  Activity measured by 5 Actical accelerometers

CONTACTS AND LOCATIONS:
Locations (1):
- Neurologic Department, Hillerød Hospital, Hillerød, Denmark